CLINICAL TRIAL: NCT05433363
Title: Renji Alzheimer's Disease Neuroimaging Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2021-260-B
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum retention in -80℃ fridge for ApoE4 gene test etc
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal control: normal, cognitive test normal, PET(-)
- cognitive disorder due to AD: PET Aβ（+），MCI-AD and AD dementia
- cognitive disorder NOT due to AD: PET Aβ（-），MCI or dementia not due to AD

SUMMARY:
This study focuses on the population of Alzheimer disease (AD). Based on Aβ(A)-Tau(T)-Vascular(V)-Neurodegeneration(N) (ATV(N))-AD evaluation system of NIA-AA Association, it can accurately diagnose and predict early AD. Positron emission tomography (PET) - magnetic resonance (MR) was used to perform Aβ、Tau molecular imaging, representing A and T in the system respectively; The quantitative detection of glucose metabolism in the brain by fluorodeoxyglucose PET (FDG-PET) can reflect the degree of neuronal damage (N); In addition, PET-MR can be used to synchronously evaluate the patients' vascular comorbidity (SVD load score) (V). Through the preliminary construction of this system, to clarify the central deposition pattern of Aβ、tau protein and the characteristics of FDG metabolism; To clarify the correlation between PET-MR imaging indexes and the progression of early cognitive impairment in AD, and to clarify the role of degeneration and vascular factors in the occurrence and development of AD; To provide a preliminary basis for the subsequent establishment of a molecular imaging model for the prognosis of early AD.

DETAILED DESCRIPTION:
Alzheimer disease (AD) is the most common cognitive impairment disease, which is mainly manifested in memory loss, language function and logical thinking disorder, and ultimately leads to the loss of independent living ability of patients. China has become the country with the largest number of AD patients in the world. At present, it has reached more than 8 million. The AD incidence rate of the elderly over 65 years old is 4%-6%, which seriously affects the health of the elderly. At present, the medicines used in clinical practice are only symptomatic treatment, and have no effect on reversing the course of disease. Studies have shown that AD has a preclinical period of more than 10 years. In this period, patients have specific pathological changes in the brain, but there are no obvious clinical symptoms. However, if the intervention is started after significant cognitive impairment, irreversible changes have taken place in the brain, and the intervention effect is limited. In recent years, many drug clinical studies on ad specific pathophysiological processes have not achieved positive results, which may be one of the important reasons why the study failed to include subjects in the early stage of the disease.

In this context, in 2011, the National Institute of Aging and the Alzheimer's Association (NIA-AA) developed diagnostic criteria for preclinical AD, mild cognitive impairment (MCI) due to AD, and dementia due to AD, which are based on AD specific biomarkers, transform the prenatal diagnosis of AD from clinical symptomatology architecture to central biomarker architecture (gold standard). The latter refers to β Amyloid protein（Aβ), Phosphorylated tau (p-tau) and secondary neurodegenerative injury (neurodegeneration), the so-called AT(N) architecture, in which "A" and "T" are AD specific lesions, and "A" is the earliest landmark change. Through in vivo detection of AD specific central markers to identify AD as early as possible and carry out targeted intervention, it is expected to provide the possibility for AD reversal. On the other hand, it is well known that AD tends to occur in the elderly, and there are often small vessel disease (SVD) coexisting in varying degrees. Both can work together to lead to AD progression. How to define the interaction between the two in the occurrence and progression of disease is also the focus of clinical research on AD. In this context, the 2018 NIA-AA standard update pointed out that the AT(N) architecture can be extended according to the AD comorbidity. For example, if AD is complicated with cerebrovascular disease, AT (N) can be correspondingly extended to ATV (N). The international clinical research based on AT(N) is very limited, while the research on ATV (N) is blank at present.

At present, PET-CT or PET-MR can be used to perform aβ and Tau molecular imaging and FDG-PET can reflect the damage degree of neurons through the quantitative detection of brain glucose metabolism, and realize the early accurate individual diagnosis of AD based on AT(N) architecture. PET-MR can also realize the simultaneous evaluation of patients' vascular comorbidity. For example, the SVD load score of MRI images is often used in clinical evaluation. Therefore, PET-MR research is carried out on patients with AD-MCI, It can realize the early accurate identification and comprehensive evaluation of AD based on AT(V) N architecture, and help to explore the contribution of degenerative factors and vascular load to the occurrence and development of cognition. It is a hot spot in clinical research in the field of AD at present, and it is in urgent need of breakthrough. At present, the research on the central biomarkers of early clinical AD is very limited, especially the longitudinal study which is combination of Aβ、 Tau and FDG multimodal PET images.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 50-75 years old; 2) complaints of memory decline; 3) Education≥ 6 years; 4) Be able to cooperate with the whole neuropsychological examinations; 5) No PET-MRI or brain MRI contraindications; 6) Sign informed consent.
* normal control: 1) Age: 50-75 years old; 2) No complaints of memory decline; 3) Mini-Mental State Examination (MMSE) ≥ 26 points; 4) Education years ≥ 6 years; 5) Be able to cooperate with a full set of neuropsychological examinations; 6) No PET-MRI or brain MRI contraindications; 7) Sign informed consent.

Exclusion Criteria:

* 1) Serious mental illness; 2) Severe depression: Hamilton Depression Scale (HAMD-17) scores ≥ 24; 3) Serious heart, liver, kidney and other important organ diseases; 4) PET-MRI or brain MRI contraindications

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care population; primary care clinic; memory clinic
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
To establish AD accurate evaluation model | from 2022-02 to 2022-08
  Using PET-MR to establish AD accurate evaluation model based on ATV (N) evaluation system
to analyze the correlation of PET-MR imaging indicators in AD progression | From 2022-08 to 2023-02
  PET-MR imaging indicators were used to analyze the correlation between the progress of cognitive impairment in AD and to prepare for the follow-up study
To clarify the role of degeneration and vascular factors in the development of cognition | From 2022-08 to 2023-02
  To clarify the role of degeneration and vascular factors in the development of cognition

CONTACTS AND LOCATIONS:
Overall Officials: Qun Xu, professor, Principal Investigator — Renji Hospital, Shanghai Jiaotong University of Medicine
Locations (1):
- Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dubois B, Feldman HH, Jacova C, Cummings JL, Dekosky ST, Barberger-Gateau P, Delacourte A, Frisoni G, Fox NC, Galasko D, Gauthier S, Hampel H, Jicha GA, Meguro K, O'Brien J, Pasquier F, Robert P, Rossor M, Salloway S, Sarazin M, de Souza LC, Stern Y, Visser PJ, Scheltens P. Revising the definition of Alzheimer's disease: a new lexicon. Lancet Neurol. 2010 Nov;9(11):1118-27. doi: 10.1016/S1474-4422(10)70223-4. Epub 2010 Oct 9. PMID 20934914
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Visser PJ, Tijms B. Brain Amyloid Pathology and Cognitive Function: Alzheimer Disease Without Dementia? JAMA. 2017 Jun 13;317(22):2285-2287. doi: 10.1001/jama.2017.6895. No abstract available. PMID 28609518
- [Background] Jack CR Jr, Albert MS, Knopman DS, McKhann GM, Sperling RA, Carrillo MC, Thies B, Phelps CH. Introduction to the recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):257-62. doi: 10.1016/j.jalz.2011.03.004. Epub 2011 Apr 21. PMID 21514247
- [Background] Pantoni L, Gorelick P. Advances in vascular cognitive impairment 2010. Stroke. 2011 Feb;42(2):291-3. doi: 10.1161/STROKEAHA.110.605097. Epub 2011 Jan 13. No abstract available. PMID 21233478
- [Background] Dichgans M, Leys D. Vascular Cognitive Impairment. Circ Res. 2017 Feb 3;120(3):573-591. doi: 10.1161/CIRCRESAHA.116.308426. PMID 28154105
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Anderson ND. State of the science on mild cognitive impairment (MCI). CNS Spectr. 2019 Feb;24(1):78-87. doi: 10.1017/S1092852918001347. Epub 2019 Jan 17. PMID 30651152
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Farias ST, Mungas D, Reed BR, Harvey D, DeCarli C. Progression of mild cognitive impairment to dementia in clinic- vs community-based cohorts. Arch Neurol. 2009 Sep;66(9):1151-7. doi: 10.1001/archneurol.2009.106. PMID 19752306
- [Background] Tolar M, Abushakra S, Hey JA, Porsteinsson A, Sabbagh M. Aducanumab, gantenerumab, BAN2401, and ALZ-801-the first wave of amyloid-targeting drugs for Alzheimer's disease with potential for near term approval. Alzheimers Res Ther. 2020 Aug 12;12(1):95. doi: 10.1186/s13195-020-00663-w. PMID 32787971
- [Background] Staals J, Booth T, Morris Z, Bastin ME, Gow AJ, Corley J, Redmond P, Starr JM, Deary IJ, Wardlaw JM. Total MRI load of cerebral small vessel disease and cognitive ability in older people. Neurobiol Aging. 2015 Oct;36(10):2806-11. doi: 10.1016/j.neurobiolaging.2015.06.024. Epub 2015 Jun 26. PMID 26189091
- [Background] Staals J, Makin SD, Doubal FN, Dennis MS, Wardlaw JM. Stroke subtype, vascular risk factors, and total MRI brain small-vessel disease burden. Neurology. 2014 Sep 30;83(14):1228-34. doi: 10.1212/WNL.0000000000000837. Epub 2014 Aug 27. PMID 25165388
- [Background] Jessen F, Amariglio RE, Buckley RF, van der Flier WM, Han Y, Molinuevo JL, Rabin L, Rentz DM, Rodriguez-Gomez O, Saykin AJ, Sikkes SAM, Smart CM, Wolfsgruber S, Wagner M. The characterisation of subjective cognitive decline. Lancet Neurol. 2020 Mar;19(3):271-278. doi: 10.1016/S1474-4422(19)30368-0. Epub 2020 Jan 17. PMID 31958406